CLINICAL TRIAL: NCT00942175
Title: A Phase 1, Randomized, Open-Label, 2-Period, Crossover Design Study to Assess the Effects of Multiple Oral Doses of Dexlansoprazole, Lansoprazole, Omeprazole or Esomeprazole on the Steady-State Pharmacokinetics and Pharmacodynamics of Clopidogrel in Healthy Subjects
Brief Title: A Study of the Effects of Multiple Doses of Dexlansoprazole, Lansoprazole, Omeprazole or Esomeprazole on the Pharmacokinetics and Pharmacodynamics of Clopidogrel in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: TAK-390MR_101; U1111-1112-6792 (Registry Identifier: WHO)
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Results first posted 2011-09-07 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Pharmacology; Stomach Ulcer; Esophagitis, Peptic; Zollinger-Ellison Syndrome; Platelet function; PPI; clopidogrel; Pharmacokinetics and Pharmacodynamics
MeSH Terms: conditions — Stomach Ulcer; Esophagitis, Peptic; Zollinger-Ellison Syndrome | interventions — Clopidogrel; Lansoprazole; Dexlansoprazole; Omeprazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Regimen A (Other): Clopidogrel 75 mg QD
  Interventions: Drug: Clopidogrel
- Regimen B (Other): Clopidogrel 75 mg QD and Lansoprazole 30 mg QD
  Interventions: Drug: Clopidogrel and Lansoprazole
- Regimen C (Other): Clopidogrel 75 mg QD and Dexlansoprazole 60 mg QD
  Interventions: Drug: Clopidogrel and Dexlansoprazole
- Regimen D (Other): Clopidogrel 75 mg QD and Omeprazole 80 mg QD
  Interventions: Drug: Clopidogrel and Omeprazole
- Regimen E (Other): Clopidogrel 75 mg QD and Esomeprazole 40 mg QD
  Interventions: Drug: Clopidogrel and Esomeprazole

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg, tablets, orally, once daily days 1-9.
  Other Names: Plavix
  Arms: Regimen A
Drug: Clopidogrel and Lansoprazole — Clopidogrel 75 mg, tablets, orally, once daily and Lansoprazole 30 mg, capsules, orally, once daily days 1-9.
  Other Names: Plavix; Prevacid; AG-1749
  Arms: Regimen B
Drug: Clopidogrel and Dexlansoprazole — Clopidogrel 75 mg, tablets, orally, once daily and Dexlansoprazole 60 mg, capsules, orally, once daily days 1-9.
  Other Names: Plavix; Kapidex; TAK-390MR
  Arms: Regimen C
Drug: Clopidogrel and Omeprazole — Clopidogrel 75 mg, tablets, orally, once daily and Omeprazole 80 mg, capsules, orally, once daily days 1-9.
  Other Names: Plavix
  Arms: Regimen D
Drug: Clopidogrel and Esomeprazole — Clopidogrel 75 mg, tablets, orally, once daily and Esomeprazole 40 mg, capsules, orally, once daily days 1-9.
  Other Names: Plavix; Nexium
  Arms: Regimen E

SUMMARY:
The purpose of this study is to assess the potential effect and safety of multiple oral doses of dexlansoprazole, lansoprazole, omeprazole or esomeprazole, once daily (QD), on the steady-state pharmacokinetics and pharmacodynamics of clopidogrel, and to assess the safety of multiple doses of clopidogrel in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open-label, single-center, multiple-dose, 2-period, crossover study to assess the effects of multiple oral doses of dexlansoprazole, lansoprazole, omeprazole or esomeprazole on the steady-state pharmacokinetics (PK) and pharmacodynamics (PD) of clopidogrel in healthy participants.

Participants were randomized equally into eight regimen sequence groups, 20 participants each. Participants randomized to Sequence Groups 1 and 2, 3 and 4, 5 and 6 and 7 and 8 were called proton pump inhibitor (PPI) Groups 1, 2, 3, and 4, respectively. Each sequence group consists of 2 regimens. Sequence Groups 1, 3, 5 and 7 dosed Regimen A (75 mg clopidogrel) for Days 1-9 of Period 1 and then crossed over to one of the following 4 regimens for Days 1-9 of Period 2: Regimen B (75 mg clopidogrel + 30 mg lansoprazole), Regimen C (75 mg clopidogrel + 60 mg dexlansoprazole), Regimen D (75 mg clopidogrel + 80 mg [2x40 mg] omeprazole), or Regimen E (75 mg clopidogrel + 40 mg esomeprazole). Sequence Groups 2, 4, 6 and 8 began with either Regimen B, C, D or E for Period 1 and then crossed over to Regimen A for Period 2.

On Day 9 of each period, blood samples were collected at predose and for 24 hours postdose to measure plasma concentrations of the active metabolite of clopidogrel. Platelet function was assessed daily prior to the dose of clopidogrel on Days 7-9 and 24-hours post Day 9 dose in each period. There was a washout interval of 10 to 14 days between the last dose of study drug in Period 1 and the first dose of study drug in Period 2.

Study participants were confined to the study center for 10 consecutive nights in Period 1, followed by a 10- to 14-day washout interval and confined for an additional 10 consecutive nights in Period 2.

ELIGIBILITY:
Inclusion Criteria:

1. The participant or the participant's legally acceptable representative signs a written, informed consent form prior to the initiation of any study procedures.
2. Weighs at least 50 kg and has a body mass index (BMI) between 18 and 30 kg/m2, inclusive, at Screening and Check-in (Day -1 of Period 1) Visits.
3. Must be a CYP2C19 extensive metabolizer (wt/wt).
4. Females cannot be nursing and must have a negative urine pregnancy test at Day -1 or be of non-childbearing potential. If females are of child bearing potential, must have a negative serum human chorionic gonadotropin (hCG) pregnancy test during Screening and on an acceptable form of contraception, or have had bilateral tubal ligation if performed a minimum of 90 days prior to Day 1.
5. At the Screening and Check-in (Day -1 of Period 1) Visits, must have an estimated creatinine clearance (CLcr) greater than or equal 90 mL/minute as determined from the Cockcroft-Gault formula.
6. Is in good health as determined by a physician based upon medical history, electrocardiogram, and physical examination findings at the Screening and Check-in (Day -1 of Period 1) Visits.
7. Participant's clinical laboratory evaluations (including hematology, clinical chemistry [fasted for a least 8 hours], and urinalysis) at the Screening and Check-in (Day -1 of Period 1) Visits are within the reference range for the testing laboratory or are deemed not clinically significant by the investigator and TGRD Medical Monitor.
8. Participant's urine drug screen for selected substances of abuse is negative at the Screening and Check-in (Day -1 of Period 1) Visits.

Exclusion Criteria:

1. Has consumed products containing Seville oranges (sour), grapefruit or grapefruit juice within 14 days prior to the first dose of study drug or is unwilling to agree to abstain from products containing Seville oranges (sour), grapefruit or grapefruit juice while participating in the study.
2. Has current or recent (within 6 months) gastrointestinal disease, a history of malabsorption, esophageal reflux, gastric bleeding or peptic ulcer disease, frequent (more than once per week) occurrence of heartburn, or any surgical intervention (eg, cholecystectomy), which would be expected to influence the absorption of drugs.
3. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as the consumption of more than 4 alcoholic beverages per day) within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
4. Is currently participating in another investigational study or has received any investigational compound within 30 days prior to the Check-in (Day -1 of Period 1) Visit.
5. Has received any known hepatic or renal clearance altering agents (eg, erythromycin, cimetidine, barbiturates, phenothiazines, fluvoxamine, etc.) within 28 days prior to first dose of study drug.
6. Has a history or clinical manifestations of significant metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urologic, immunologic, or psychiatric disorder as determined by the investigator which may impact the ability of the participant to take part in or potentially confound the trial results.
7. Has a history of hypersensitivity or allergies to any drug or food or any excipients of clopidogrel, lansoprazole, dexlansoprazole, omeprazole, esomeprazole or other drug with the same mechanism of action or related compounds.
8. Has had an acute, clinically significant illness within 30 days prior to the first dose of study drug.
9. Has a systolic blood pressure greater than 140 mm Hg or has a diastolic blood pressure greater than 90 mm Hg at Screening or Check-in (Day -1 of Period 1).
10. Has a positive test result for hepatitis B surface antigen (HBsAg) or antibody to hepatitis C virus (anti-HCV) at Screening, or a known history of infection with the human immunodeficiency virus (HIV).
11. Has a Day -1 laboratory value assessed by the principal investigator and sponsor medical monitor as clinically significant underlying disease or condition that may prevent the participant from entering the study.
12. Has an alanine aminotransferase, aspartate aminotransferase or Total Bilirubin level that exceeds the upper limit of normal at the Screening or Check-in (Day -1 of Period 1) Visits.
13. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 6 weeks prior to Check-in (Day -1 of Period 1) Visit, or has a positive cotinine screen at the Screening or Check-in (Day - 1 of Period 1) Visits or anticipates an inability to abstain from these products for the duration of the study.
14. With the exception of acetaminophen, has taken any excluded medication, supplements or food products listed in the Excluded Dietary Items and Medications table located in the study protocol.
15. Has donated blood products (such as plasma) within 30 days, or has donated whole blood or had a significant blood loss (500 mL) within 56 days of the first dose of study drug
16. Has a positive test result for caffeine at the Check-in (Day -1 of Period 1) Visit.
17. Has a history of cancer, except basal cell carcinoma, which has not been in remission for at least 5 years prior to the first dose of study drug.
18. Has received clopidogrel or any PPIs or histamine2-receptor antagonists within 28 days of screening.
19. Participant, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Tempe, Arizona, United States

REFERENCES:
- [Derived] Frelinger AL 3rd, Bhatt DL, Lee RD, Mulford DJ, Wu J, Nudurupati S, Nigam A, Lampa M, Brooks JK, Barnard MR, Michelson AD. Clopidogrel pharmacokinetics and pharmacodynamics vary widely despite exclusion or control of polymorphisms (CYP2C19, ABCB1, PON1), noncompliance, diet, smoking, co-medications (including proton pump inhibitors), and pre-existent variability in platelet function. J Am Coll Cardiol. 2013 Feb 26;61(8):872-9. doi: 10.1016/j.jacc.2012.11.040. Epub 2013 Jan 16. PMID 23333143
- [Derived] Frelinger AL 3rd, Lee RD, Mulford DJ, Wu J, Nudurupati S, Nigam A, Brooks JK, Bhatt DL, Michelson AD. A randomized, 2-period, crossover design study to assess the effects of dexlansoprazole, lansoprazole, esomeprazole, and omeprazole on the steady-state pharmacokinetics and pharmacodynamics of clopidogrel in healthy volunteers. J Am Coll Cardiol. 2012 Apr 3;59(14):1304-11. doi: 10.1016/j.jacc.2011.12.024. PMID 22464259
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at one site in the United States from 15 December 2009 to 08 July 2010.
Pre-assignment Details: Healthy participants were enrolled in one of 4, once-daily (QD), proton pump inhibitor (PPI) treatment groups.
Groups:
- PPI Group 1: Regimen A: Clopidogrel 75 mg, tablets, orally, once daily for up to 9 days.
  Regimen B: Clopidogrel 75 mg, tablets, orally, once daily and Lansoprazole 30 mg, capsules, orally, once daily for up to 9 days.
- PPI Group 2: Regimen A: Clopidogrel 75 mg, tablets, orally, once daily for up to 9 days.
  Regimen C: Clopidogrel 75 mg, tablets, orally, once daily and Dexlansoprazole 60 mg, capsules, orally, once daily for up to 9 days.
- PPI Group 3: Regimen A: Clopidogrel 75 mg, tablets, orally, once daily for up to 9 days.
  Regimen D: Clopidogrel 75 mg, tablets, orally, once daily and Omeprazole 80 mg, capsules, orally, once daily for up to 9 days.
- PPI Group 4: Regimen A: Clopidogrel 75 mg, tablets, orally, once daily for up to 9 days.
  Regimen E: Clopidogrel 75 mg, tablets, orally, once daily and Esomeprazole 40 mg, capsules, orally, once daily for up to 9 days.
Period: Overall Study
Arm/Group | PPI Group 1 | PPI Group 2 | PPI Group 3 | PPI Group 4
Started | 40 | 40 | 40 | 40
Completed | 38 | 36 | 38 | 38
Not Completed | 2 | 4 | 2 | 2
Not completed — Adverse Event | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 2 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Elevated Alanine Amino Transferase | 0 | 0 | 0 | 1
Not completed — Low Platelet Count | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PPI Group 1 | PPI Group 2 | PPI Group 3 | PPI Group 4 | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 160
Age Continuous [Mean (Standard Deviation); unit: years] | 32.8 (6.48) | 35.7 (7.92) | 34.0 (7.40) | 33.3 (7.10) | 33.9 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 20 | 80
  Male | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter Peak Plasma Concentration (Cmax) of Clopidogrel's Active Metabolite.
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 9 of each period
Population: All participants who had valid parameter estimates for both regimens within a PPI group were included in the pharmacokinetics (PK) statistical analyses for this parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PPI Group 1: Regimen A; PPI Group 2: Regimen A; PPI Group 3: Regimen A; PPI Group 4: Regimen A: Clopidogrel 75 mg, tablets, orally, once daily for up to 9 days.
- PPI Group 1: Regimen B: Clopidogrel 75 mg, tablets, orally, once daily and Lansoprazole 30 mg, capsules, orally, once daily for up to 9 days.
- PPI Group 2: Regimen C: Clopidogrel 75 mg, tablets, orally, once daily and Dexlansoprazole 60 mg, capsules, orally, once daily for up to 9 days.
- PPI Group 3: Regimen D: Clopidogrel 75 mg, tablets, orally, once daily and Omeprazole 80 mg, capsules, orally, once daily for up to 9 days.
- PPI Group 4: Regimen E: Clopidogrel 75 mg, tablets, orally, once daily and Esomeprazole 40 mg, capsules, orally, once daily for up to 9 days.
Arm/Group | PPI Group 1: Regimen A | PPI Group 1: Regimen B | PPI Group 2: Regimen A | PPI Group 2: Regimen C | PPI Group 3: Regimen A | PPI Group 3: Regimen D | PPI Group 4: Regimen A | PPI Group 4: Regimen E
Number analyzed (Participants) | 38 | 38 | 36 | 36 | 38 | 38 | 38 | 38
ng/mL | 39.14 (12.553) | 30.01 (15.264) | 38.85 (15.699) | 29.33 (12.400) | 38.25 (12.461) | 22.55 (10.682) | 40.98 (22.908) | 24.69 (10.641)
Statistical Analysis 1: Comparison: PPI Group 1: Regimen A vs PPI Group 1: Regimen B; Test type: Superiority or Other; Mean Difference (Final Values) = 0.7000, 90% CI 2-sided [0.6106 to 0.8026] — The mean difference refers to the point estimates of the relative bioavailability. With its confidence intervals, it was obtained from the ANOVA model on the natural logarithm transformed data
Statistical Analysis 2: Comparison: PPI Group 2: Regimen A vs PPI Group 2: Regimen C; Test type: Superiority or Other; Mean Difference (Final Values) = 0.7340, 90% CI 2-sided [0.6516 to 0.8269] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PPI Group 3: Regimen A vs PPI Group 3: Regimen D; Test type: Superiority or Other; Mean Difference (Final Values) = 0.5564, 90% CI 2-sided [0.4877 to 0.6347] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PPI Group 4: Regimen A vs PPI Group 4: Regimen E; Test type: Superiority or Other; Mean Difference (Final Values) = 0.6783, 90% CI 2-sided [0.5063 to 0.9087] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Pharmacokinetic Parameter Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]) of Clopidogrel's Active Metabolite.
Description: Area under the plasma concentration versus time curve (AUC(0-tlqc)) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: Day 9 of each period
Population: All participants who had valid parameter estimates for both formulations within PPI groups were included in the PK statistical analyses for those parameters.
Measure: Mean (Standard Deviation); unit: ng*hr/ML
Arm/Group | PPI Group 1: Regimen A | PPI Group 1: Regimen B | PPI Group 2: Regimen A | PPI Group 2: Regimen C | PPI Group 3: Regimen A | PPI Group 3: Regimen D | PPI Group 4: Regimen A | PPI Group 4: Regimen E
Number analyzed (Participants) | 38 | 38 | 36 | 36 | 38 | 38 | 38 | 38
ng*hr/ML | 41.69 (10.020) | 36.42 (10.825) | 41.25 (14.690) | 37.75 (13.132) | 37.78 (12.043) | 26.28 (8.800) | 42.35 (18.785) | 31.23 (9.938)
Statistical Analysis 1: Comparison: PPI Group 1: Regimen A vs PPI Group 1: Regimen B; Test type: Superiority or Other; Mean Difference (Final Values) = 0.8573, 90% CI 2-sided [0.8020 to 0.9165] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PPI Group 2: Regimen A vs PPI Group 2: Regimen C; Test type: Superiority or Other; Mean Difference (Final Values) = 0.9103, 90% CI 2-sided [0.8567 to 0.9672] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PPI Group 3: Regimen A vs PPI Group 3: Regimen D; Test type: Superiority or Other; Mean Difference (Final Values) = 0.6943, 90% CI 2-sided [0.6438 to 0.7487] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PPI Group 4: Regimen A vs PPI Group 4: Regimen E; Test type: Superiority or Other; Mean Difference (Final Values) = 0.8389, 90% CI 2-sided [0.6440 to 1.0928] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Pharmacodynamic Parameter Platelet Reactivity Index (PRI) From Vasodilator-stimulated Phosphoprotein (VASP) Phosphorylation State (Flow Cytometry).
Description: PRI is the platelet reactivity index from VASP phosphorylation state (flow cytometry).
Time Frame: 24-hour post Day 9 dose in each period.
Population: All participants who had valid parameter estimates for both regimens within a PPI group were included in the pharmacodynamics (PD) statistical analyses for this parameter.
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | PPI Group 1: Regimen A | PPI Group 1: Regimen B | PPI Group 2: Regimen A | PPI Group 2: Regimen C | PPI Group 3: Regimen A | PPI Group 3: Regimen D | PPI Group 4: Regimen A | PPI Group 4: Regimen E
Number analyzed (Participants) | 38 | 38 | 36 | 36 | 38 | 38 | 38 | 38
percent inhibition | 42.3 (14.61) | 46.4 (16.44) | 41.3 (15.45) | 43.0 (16.47) | 47.9 (15.70) | 59.1 (17.87) | 46.5 (17.28) | 58.0 (14.64)
Statistical Analysis 1: Comparison: PPI Group 1: Regimen A vs PPI Group 1: Regimen B; Test type: Superiority or Other; Mean Difference (Final Values) = 4.1016, 90% CI 2-sided [0.0348 to 8.1684] — Included only participants with complete data for both regimens. Values are least squares mean difference
Statistical Analysis 2: Comparison: PPI Group 2: Regimen A vs PPI Group 2: Regimen C; Test type: Superiority or Other; Mean Difference (Final Values) = 2.0474, 90% CI 2-sided [-0.8555 to 4.9503] — Included only participants with complete data for both regimens. Values are least squares mean difference
Statistical Analysis 3: Comparison: PPI Group 3: Regimen A vs PPI Group 3: Regimen D; Test type: Superiority or Other; Mean Difference (Final Values) = 11.0407, 90% CI 2-sided [6.5219 to 15.5595] — Included only participants with complete data for both regimens. Values are least squares mean difference
Statistical Analysis 4: Comparison: PPI Group 4: Regimen A vs PPI Group 4: Regimen E; Test type: Superiority or Other; Mean Difference (Final Values) = 11.4437, 90% CI 2-sided [7.1791 to 15.7083] — Included only participants with complete data for both regimens. Values are least squares mean difference

4. Primary Outcome: Pharmacodynamic Parameter Maximum Platelet Aggregation (MPA) From Aggregometry (Turbidimetric) With 5 µM Adenosine Diphosphate.
Description: Maximum platelet aggregation (MPA) from aggregometry (turbidimetric) with 5 µM adenosine diphosphate.
Time Frame: 24-hour post Day 9 dose in each period.
Population: All participants who had valid parameter estimates for both formulations within PPI groups were included in the PD statistical analyses for those parameters.
Measure: Mean (Standard Deviation); unit: percentage of MPA
Arm/Group | PPI Group 1: Regimen A | PPI Group 1: Regimen B | PPI Group 2: Regimen A | PPI Group 2: Regimen C | PPI Group 3: Regimen A | PPI Group 3: Regimen D | PPI Group 4: Regimen A | PPI Group 4: Regimen E
Number analyzed (Participants) | 38 | 38 | 36 | 36 | 37 | 37 | 38 | 38
percentage of MPA | 28.1 (6.76) | 30.8 (9.35) | 34.6 (14.23) | 36.2 (16.87) | 34.2 (12.32) | 42.5 (14.74) | 29.3 (10.41) | 38.2 (17.77)
Statistical Analysis 1: Comparison: PPI Group 1: Regimen A vs PPI Group 1: Regimen B; Test type: Superiority or Other; p = 0.035, ANOVA — From ANOVA models in which the least-square means between two regimens are compared
Statistical Analysis 2: Comparison: PPI Group 2: Regimen A vs PPI Group 2: Regimen C; Test type: Superiority or Other; p = 0.445, ANOVA — From ANOVA models in which the least-square means between two regimens are compared
Statistical Analysis 3: Comparison: PPI Group 3: Regimen A vs PPI Group 3: Regimen D; Test type: Superiority or Other; p < 0.001, ANOVA — From ANOVA models in which the least-square means between two regimens are compared
Statistical Analysis 4: Comparison: PPI Group 4: Regimen A vs PPI Group 4: Regimen E; Test type: Superiority or Other; p < 0.001, ANOVA — From ANOVA models in which the least-square means between two regimens are compared

5. Primary Outcome: Pharmacodynamic Parameter MPA From Aggregometry (Turbidimetric) With 20 µM Adenosine Diphosphate.
Description: MPA from aggregometry (turbidimetric) with 20 µM adenosine diphosphate.
Time Frame: 24-hour post Day 9 dose in each period.
Population: All participants who had valid parameter estimates for both formulations within PPI groups were included in the PK and PD statistical analyses for those parameters.
Measure: Mean (Standard Deviation); unit: percentage of MPA
Arm/Group | PPI Group 1: Regimen A | PPI Group 1: Regimen B | PPI Group 2: Regimen A | PPI Group 2: Regimen C | PPI Group 3: Regimen A | PPI Group 3: Regimen D | PPI Group 4: Regimen A | PPI Group 4: Regimen E
Number analyzed (Participants) | 38 | 38 | 36 | 36 | 37 | 37 | 38 | 38
percentage of MPA | 36.7 (9.11) | 41.6 (12.65) | 43.1 (13.24) | 46.3 (16.93) | 43.5 (14.00) | 53.5 (13.75) | 39.3 (13.22) | 47.9 (15.77)
Statistical Analysis 1: Comparison: PPI Group 1: Regimen A vs PPI Group 1: Regimen B; Test type: Superiority or Other; p = 0.004, ANOVA — From ANOVA models in which the least-square means between two regimens are compared
Statistical Analysis 2: Comparison: PPI Group 2: Regimen A vs PPI Group 2: Regimen C; Test type: Superiority or Other; p = 0.148, ANOVA — From ANOVA models in which the least-square means between two regimens are compared
Statistical Analysis 3: Comparison: PPI Group 3: Regimen A vs PPI Group 3: Regimen D; Test type: Superiority or Other; p < 0.001, ANOVA — From ANOVA models in which the least-square means between two regimens are compared
Statistical Analysis 4: Comparison: PPI Group 4: Regimen A vs PPI Group 4: Regimen E; Test type: Superiority or Other; p < .0001, ANOVA — From ANOVA models in which the least-square means between two regimens are compared

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started or worsened after the first dose of study drug and within 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study drug.
Arm/Group | PPI Group 1: Regimen A | PPI Group 1: Regimen B | PPI Group 2: Regimen A | PPI Group 2: Regimen C | PPI Group 3: Regimen A | PPI Group 3: Regimen D | PPI Group 4: Regimen A | PPI Group 4: Regimen E
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 1/40 | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 13/39 | 16/39 | 19/39 | 16/38 | 14/40 | 11/38 | 17/39 | 15/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PPI Group 1: Regimen A (N=40) | PPI Group 1: Regimen B (N=40) | PPI Group 2: Regimen A (N=40) | PPI Group 2: Regimen C (N=40) | PPI Group 3: Regimen A (N=40) | PPI Group 3: Regimen D (N=40) | PPI Group 4: Regimen A (N=40) | PPI Group 4: Regimen E (N=40)
Serum sickness-like reaction (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PPI Group 1: Regimen A (N=39) | PPI Group 1: Regimen B (N=39) | PPI Group 2: Regimen A (N=39) | PPI Group 2: Regimen C (N=38) | PPI Group 3: Regimen A (N=40) | PPI Group 3: Regimen D (N=38) | PPI Group 4: Regimen A (N=39) | PPI Group 4: Regimen E (N=39)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 3 | 5 | 1 | 1 | 0 | 0 | 1
Feeling Hot (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1 | 2 | 1 | 2 | 0
Headache (Nervous system disorders) | 3 | 4 | 5 | 7 | 2 | 6 | 6 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 3 | 4 | 2 | 2 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 3 | 1 | 0 | 2 | 2
Somnolence (Nervous system disorders) | 1 | 1 | 2 | 1 | 1 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 2 | 0 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 3 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights therefrom or any data, information or materials obtained or generated in the performance of it's obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.